CLINICAL TRIAL: NCT04812912
Title: The Effects of Chemotherapy or Radiotherapy on Reproductive and Sexual Health of Early Onset Colorectal Cancer Patients
Brief Title: Changes in Reproductive and Sexual Health in People With Early Onset Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-035
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Carcinoma
Keywords: Early Onset Colorectal Cancer; Colorectal Cancer; 21-035; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Colon Cancer: This patient population will have hormone biomarker analysis, questionnaire (QOL) administration, and, if the patient is male, semen analysis
  Interventions: Diagnostic Test: Hormone biomarker analysis; Behavioral: QoL Questionnaires
- Participants with Rectal Cancer: This patient population will have hormone biomarker analysis, QOL administration, and, if the patient is male, semen analysis
  Interventions: Diagnostic Test: Hormone biomarker analysis; Behavioral: QoL Questionnaires

INTERVENTIONS:
Diagnostic Test: Hormone biomarker analysis — For female patients, hormone biomarker analysis will be performed to measure: anti-Mullerian hormone (AMH), estradiol and FSH in the blood. In male patients, hormone biomarkers of testicular function and spermatogenesis will be monitored: testosterone, inhibin B, steroid hormone binding globulin (SHBG) and FSH. Sperm analysis will also be performed in male patients to monitor changes in sperm count.
Behavioral: QoL Questionnaires — All participants will respond to protocol questionnaires, which will include both validated questionnaires as well as non-validated ones. This design will allow for basic demographic, psychosocial and sexual-health-related data to be obtained.

SUMMARY:
The purpose of this study is to find out how cancer treatments (chemotherapy and/or radiation therapy) affect reproductive and sexual health in people with early onset colorectal cancer. The study researchers will observe and track changes in hormone levels and in sexual and reproductive health in people with early onset colorectal cancer. This information will help researchers know more about how cancer treatments affect reproductive and sexual health, including the ability to have children (fertility).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age and premenopausal (female) or 18-50 years of age (male) at time of diagnosis
* Histologic diagnosis of colorectal adenocarcinoma
* Able and willing to participate in the informed consent process
* Eligible for curative adjuvant or neoadjuvant therapy for colon or rectal cancer
* Willing and able to complete protocol questionnaires
* Rectal patients only: Individuals who will be receiving chemotherapy, followed by chemoradiotherapy (ChemoRT)

Exclusion Criteria:

* Prior systemic treatment for this malignancy
* Active or prior secondary malignancy
* History of ovarian resection (if female)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception until the termination of gestation, confirmed by a positive hCG laboratory test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential research subjects will be identified through the Center for Young Onset Colorectal Cancer, a member of the patient's treatment team, the principal investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC). All study participants will be recruited from patients under the care of consenting professionals. If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Change in anti-Mullerian hormone (AMH), estradiol and FSH of oxaliplatin-induced gonadal toxicity in pre-menopausal female patients (<40y) | Up to 30 months
Change in testosterone, inhibin B, steroid hormone binding globulin (SHBG) and FSH in young male patients (<50y) undergoing therapy for colorectal cancer | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org